CLINICAL TRIAL: NCT03482960
Title: Comparison of 129Xe MRI With 19F MRI in CF Lung Disease
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 17-2569; XePFP2017 (Other: University of North Carolina at Chapel Hill)
Record Dates: First submitted 2018-03-23; First posted 2018-03-29 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2020-09

CONDITIONS: Cystic Fibrosis
Keywords: imaging; hyperpolarized; perfluorinated; MRI; lung
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 129Xe MRI (Experimental): Participants will self-administer hyperpolarized xenon gas via inhalation prior to the investigators acquiring MRI images. MRI imaging will be taken during approximately 15-second breath-holds. After the MRI is complete, participant performs spirometry maneuvers in a room outside the magnet. Once a minimum of 15 minutes has elapsed since leaving the MRI scanner, the participant will return to the MRI scanner, where the second phase of the study will occur. PFP gas will be administered using a full-face mask during the MRI. Images are acquired during 12-second breath-hold after every 3rd breath.
  Interventions: Drug: Hyperpolarized Xenon gas; Drug: PFP
- 19F MRI with PFP (Experimental): PFP gas will be administered using a full-face mask during the MRI. Images are acquired during 12-second breath-hold after every 3rd breath. After the MRI is complete, participant performs spirometry maneuvers in a room outside the magnet. Once a minimum of 15 minutes has elapsed since leaving the MRI scanner, the participant returns to the MRI scanner, where he/she will self-administer hyperpolarized xenon gas prior to acquiring MRI images. MRI imaging will be taken during approximately 15-second breath-holds.
  Interventions: Drug: Hyperpolarized Xenon gas; Drug: PFP

INTERVENTIONS:
Drug: Hyperpolarized Xenon gas — Hyperpolarized Xenon gas
  * Hyperpolarized mixture (750ml HP 129Xe and 250ml nitrogen)
  * Administration: By mouthpiece attached to a single use Tedlar bag.
  * Dosage: 750 mL of the 129Xe mixture up to, but not exceeding, four doses of the 129Xe.
  * Frequency: 10-minute interval between doses.
  Other Names: 129Xe
Drug: PFP — * Inhaled PFP, a gaseous contrast agent (79% PFP; 21% O2, pre-mixed, medical grade gas)
  * Administration: Full-face disposable ventilation mask and a standard Douglas Bag system.
  * Dosage: Two controlled breaths of the contrast gas followed by a full breath and a 12-second breath-hold and scan for image acquisition.
  * Frequency: Repeated 5 times followed by an identical five cycles with room air to ensure PFP gas wash-out has occurred.
  Other Names: Perfluoropropane gas (C3F8); 19F

SUMMARY:
This study is designed to compare the capabilities of two novel imaging techniques: polarized perfluorinated gas mixed with oxygen, and hyperpolarized xenon mixed with N2 to detect changes in lung ventilation using MRI.

DETAILED DESCRIPTION:
The goal of this study is to compare the capabilities of two novel imaging techniques: conventional 'thermally' polarized perfluorinated gases (perfluoropropane, or PFP) mixed with oxygen, and hyperpolarized xenon (129Xe) mixed with N2 to detect changes in lung ventilation using magnetic resonance imaging (MRI). Although considerable work has been done internationally with hyperpolarized xenon MRI, the low availability and high cost of this technique is limiting. Perfluorinated gas MRI is an alternative that may in fact be a suitable, simpler alternative. PFP is commercially availability in large quantities, which allows multiple breath studies and thus provides the ability to analyze gas wash-in and wash-out kinetics. These endpoints may improve the investigators ability to detect ventilation abnormalities beyond the traditional "ventilation defect percentage" parameter obtained with 129Xe MRI. The commercial availability of PFP and lack of need for onsite hyperpolarization may also facilitate the transfer of this technology to other centers for the conduct of multicenter studies. The investigators hypothesize that 19F MRI will not be inferior to hyperpolarized xenon MRI in detection of ventilation defect percentages (VDP).

ELIGIBILITY:
Inclusion Criteria:

Subjects with CF must meet all of the following inclusion criteria to be eligible for enrollment:

1. Subjects must be at least 18 years of age;
2. Non-smokers (<10 pack year history and no active smoking in the past year);
3. Diagnosis of cystic fibrosis as via standard sweat chloride/phenotypic features/genotyping
4. Stable lung disease as evidenced by no change in respiratory medications or change in forced expiratory volume in 1 second (FEV1) of >15% from baseline over the preceding 4 weeks prior to enrollment
5. Baseline FEV1 >70% of predicted.
6. No use of supplemental oxygen
7. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the trial
8. Subjects must be willing and able to comply with scheduled visits and other trial procedures.

Subjects without CF must meet all of the following inclusion criteria to be eligible for enrollment:

1. Subjects must be at least 18 years of age;
2. Non-smokers (<10 pack year history and no active smoking in the past year);
3. Baseline FEV1 >70% of predicted.
4. No use of supplemental oxygen or clinically significant lung disease
5. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the trial
6. Subjects must be willing and able to comply with scheduled visits and other trial procedures.

Exclusion Criteria:

1. Active or past smokers with less than 1 years since quitting or >10 pack-year smoking history
2. Co-existent asthma (as evidenced by either clinical diagnosis, chronic oral steroid use, or marked broncho-reactivity on pulmonary function testing)
3. Unable to undergo a 3.0-Tesla MRI exam of the lungs and chest because of contraindications including

   * Occupation (past or present) of machinist, welder, grinder;
   * Injury to the eye involving a metallic object
   * Injury to the body by a metallic object (bullet, BB, shrapnel)
   * Presence of a cardiac pacemaker or defibrillator
   * Presence of aneurysm clips
   * Presence of carotid artery vascular clamp
   * Presence of neurostimulator
   * Presence of insulin or infusion pump
   * Presence of implanted drug infusion device that is not known to be MRI compatible (i.e., was placed outside of UNCH or is older than 10 years)
   * Bone growth or fusion simulator
   * Presence of cochlear, otologic or ear implant
   * Any type of prosthesis (eye, penile, etc.)
   * Artificial limb or joint
   * Non-removable electrodes (on body, head or brain)
   * Intravascular stents, filters or coils
   * Shunt (spinal or intraventricular)
   * Swan-ganz catheter
   * Any implant held in place by a magnet
   * Transdermal delivery system (e.g. Nitro)
   * Intrauterine Device (IUD) or diaphragm
   * Tattooed makeup (eyeliner, lips, etc.) or tattoos covering >25% of body surface area
   * Body piercings (MUST BE REMOVED BEFORE MRI)
   * Any metal fragments
   * Internal pacing wires
   * Metal or wire mesh implants
   * Hearing aid (REMOVE BEFORE MRI)
   * Dentures (REMOVE BEFORE MRI)
   * Claustrophobia
4. Unable to tolerate inhalation of gas mixture
5. Any changes in medications that may affect CF lung disease in the past 14 days, including any experimental therapies
6. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or may interfere with the interpretation of trial results and, in the judgment of the investigator, would make the subject inappropriate for entry into this trial.
7. Pregnancy; women of childbearing potential must have a confirmed negative urine pregnancy test on the day of the MRI scan, prior to the MRI scan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2019-04-09 (Actual); Study Completion 2019-04-10 (Actual)

PRIMARY OUTCOMES:
Volume of unventilated lung area after a single 129Xe inhalation and after each inhalation cycle with PFP | 1 hour
  Primary comparison will be the VDP with Xenon (single breath) and after first PFP inhalation cycle (3 breaths of PFP)

SECONDARY OUTCOMES:
Signal-to-noise (SNR) of each modality | 20 minutes
  Assessment of the quality of signal achieved with each modality
Rate constant describing wash-in and wash-out of PFP | 15 minutes
  change in ventilated areas of the lung over time when administered PFP
Correlation between VDP identified by each modality and spirometry and Lung Clearance Index (LCI) | 2 hours
  Comparison of VDP to two standard metrics of lung function, spirometry and LCI

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Goralski, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McCallister A, Chung SH, Antonacci M, Z Powell M, Ceppe AS, Donaldson SH, Lee YZ, Branca RT, Goralski JL. Comparison of single breath hyperpolarized 129 Xe MRI with dynamic 19 F MRI in cystic fibrosis lung disease. Magn Reson Med. 2021 Feb;85(2):1028-1038. doi: 10.1002/mrm.28457. Epub 2020 Aug 8. PMID 32770779